CLINICAL TRIAL: NCT04647981
Title: Diagnostic Performance Evaluation Study of the Xpert® Bladder Cancer Monitor Test in the Surveillance of Patients With Non-Invasive Bladder Urothelial Carcinoma.
Brief Title: Diagnostic Performance Evaluation Study of the Xpert® Bladder Cancer Monitor Test.
Acronym: Xpert Bladder
Status: Completed | Type: Observational
Sponsor: Clinique Beau Soleil (Other)
Collaborators: Cepheid (Industry); Team Languedoc Mutualité / Nouvelles technologies (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-A03392-53
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Non-Invasive Bladder Urothelial Carcinoma; Non-Invasive Bladder Papillary Urothelial Carcinoma, Low Grade; Non-Invasive Bladder Papillary Urothelial Carcinoma, High Grade
Keywords: Bladder; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xpert® Bladder Test: A urine sample is collected before cystoscopy.
  Interventions: Other: Xpert® Bladder Cancer Monitor Test

INTERVENTIONS:
Other: Xpert® Bladder Cancer Monitor Test — The urine sample is analyzed with the Xpert® Bladder Cancer Monitor test.

SUMMARY:
Non-muscle invasive bladder tumor is a condition that can recur with a risk of progression to an infiltrating tumor of the muscle. Regular follow-up is therefore essential to detect any recurrence or progression of the disease as early as possible.

Currently, the monitoring of this type of tumor is done by cystoscopy (examination that allows visualization of the bladder wall) associated with urinary cytology (analysis of urine to detect an abnormality). These examinations have their limits, they may not detect certain types of tumors or may be painful.

To reduce the number of cystoscopies and replace urinary cytology, several urinary markers have been developed in recent years. This is the case of the Xpert® Bladder Cancer Monitor test, which is a non-invasive, in vitro diagnostic urine test dedicated to the monitoring of patients with bladder cancer.

The purpose of this study is to evaluate the diagnostic performance of the Xpert® Bladder Cancer Monitor test for the detection of bladder tumor recurrence, compared to reference tests.

DETAILED DESCRIPTION:
This study consists of a urine sample. During the participant's medical consultation with his/her urologist, for the monitoring of his/her non-invasive bladder tumor(s), a cystoscopy is performed. Before the examination, the participant gives a urine sample, which will be analyzed by the Xpert®Bladder Cancer Monitor test.

The main objective of this non-interventional monocentric study is to compare the sensitivity of the Xpert® Bladder Cancer Monitor test performed on the GeneXpert® system to the sensitivity of cytology.

The reference test is a combination of cystoscopy and histology. The algorithm is as follows: if the cystoscopy is negative, it will be considered that there is no recurrence; if the cystoscopy is positive, a biopsy of the "abnormal" area will be performed and histology will be requested. If the histology is positive, it will be considered that there is a recurrence; otherwise, it will be considered that there is no recurrence.

The gold standard is, therefore, the couple: cystoscopy +/- histology

* A cystoscopy will be considered positive if to the naked eye the urologist sees a macroscopically suspicious lesion (e.g. a budding lesion).
* If the cystoscopy is positive, the urologist will take a sample of the suspect lesion and have it analyzed by the pathologist. If the lesion analyzed has the same histology as the original lesion, it will be considered a recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a social security scheme.
* Participant has signed a form of no objection to the use of the data.
* Participant has had a transurethral resection of bladder tumor revealing non-invasive-muscle bladder tumor prior to inclusion within a maximum of 5 years from the date of diagnosis to the absence of recurrence since then.
* Participant is seen for a follow-up cystoscopy on the day of the visit.

Non-Inclusion Criteria:

* Vulnerable persons (Article L 1121-6 of the Public Health Code).
* Adults subject to legal protection or unable to express their consent (Article 1121-8 of the Public Health Code).
* Persons with a bladder tumor other than a non-invasive bladder tumor (i.e., invasive bladder cancer).
* A person who has undergone bladder tumor resection or therapy with Calmette-Guerin bacilli or with Mitomycin C less than 6 weeks (42 days) prior to inclusion.

Exclusion Criteria:

- Participant no longer wishing to participate in the study, or in the course of the study with a refusal to use the data until exit from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A person with antecedents of non-invasive bladder tumors and who has had previous transurethral resection of bladder tumor.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Compare sensitivities of the Xpert® Bladder Cancer Monitor Test and the urinary cytology test. | 12 months
  The two tests, the Xpert® Bladder Cancer Monitor and the urinary cytology, made during the follow-up of patients with non-invasive-muscle bladder tumor are compared to the gold standard, which is the reference examination: the couple cystoscopy/histology.

SECONDARY OUTCOMES:
Evaluate the diagnostic accuracy of the Xpert® Bladder Cancer Monitor test. | 12 months
  Evaluate the diagnostic accuracy of the Xpert® Bladder Cancer Monitor test for the detection of bladder tumor recurrence (stage, grade).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Trabelssi, M.D., Principal Investigator — Clinique Beau Soleil
Locations (1):
- Clinique Beau Soleil, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Qualitative monitoring for recurrence in patients previously diagnosed with bladder cancer in 90 minutes. — https://www.cepheid.com/en/tests/Oncology-Genetics/Xpert-Bladder-Cancer-Monitor